CLINICAL TRIAL: NCT06099587
Title: MIMA Pilot Study: MIcrostructure of the Medial Temporal Lobe in Early Alzheimer's Disease
Acronym: MIMA-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC23_8900_MIMA-P
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: Alzheimer disease; Mild Cognitive Impairment; Subjective cognitive decline-plus; Diffusion MRI; Microstructure; Memory
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Prospective single-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCD+ (Experimental): Patients with subjective cognitive decline-plus due to Alzheimer's disease (or "DCS" in french)
  Interventions: Diagnostic Test: high-resolution diffusion MRI
- MCI (Experimental): Patients with mild neurocognitive impairment due to Alzheimer's disease (or "TCL" in french)
  Interventions: Diagnostic Test: high-resolution diffusion MRI

INTERVENTIONS:
Diagnostic Test: high-resolution diffusion MRI — The study will combine multi-compartment models (e.g. Archer et al., 2020; Parker et al., 2020) of high-resolution diffusion MRI within medial temporal lobes regions of interest defined through the ASHS algorithm (Yushkevich et al., 2015), with theoretically driven cognitive assessment medial temporal lobes functions. The '4 mountains test' and the 'Memory entities' test will allow specific probing of hippocampal and rhinal cortices functions, respectively (Hartley et al., 2007; Besson et al., 2020).
  Other Names: Memory tests

SUMMARY:
Patients with Mild Cognitive Impairment (MCI) or Subjective Cognitive Decline (SCD) may or may not develop Alzheimer's disease (AD) dementia. Yet identifying patients at risk is crucial: delaying the onset of the disease by 5 years could reduce prevalence by 50%. To achieve this, we need affordable biomarkers combined with clinically meaningful assessment tools. Current approaches (cognition, imaging or Tau and Amyloid peptide assays) lack precision or specificity (e.g., age-related memory deficits) and involve invasive and costly procedures, sometimes inaccessible in France (e.g., the "AT(N)" framework). Recently, quantitative diffusion MRI (dMRI) has identified in-vivo gray matter microstructural changes linked to hyperphosphorylated Tau protein, which are of great diagnostic value. Still, we ignore whether and how these changes are responsible for early memory impairment in AD. The MIMA-P project will combine multi-compartment models of the high-resolution diffusion signal with a cognitive assessment of memory based on recent models of medial temporal lobe function to assess the relevance of a new affordable, rapid and non-invasive early marker of the disease.

DETAILED DESCRIPTION:
The study will combine multi-compartment models (e.g. Archer et al., 2020; Parker et al., 2020) of high-resolution diffusion MRI within medial temporal lobes regions of interest defined through the ASHS algorithm (Yushkevich et al., 2015), with theoretically driven cognitive assessment medial temporal lobes functions. The '4 mountains test' and the 'Memory entities' test will allow specific probing of hippocampal and rhinal cortices functions, respectively (Hartley et al., 2007; Besson et al., 2020).

25 patients with 'subjective cognitive decline-plus' (hereafter 'SCD', criteria of Jessen et al., 2014) and 25 patients with mild neurocognitive impairment due to Alzheimer's disease (hereafter 'MCI', criteria of Albert et al., 2011) matched for gender, socio-professional category and level of education. The 25 healthy volunteers required have already been included in a different study.

ELIGIBILITY:
Inclusion Criteria:

* aged between 50 and 80
* native French speaking
* right-handed
* with a level of education equal to or higher than the Certificat d'Etudes Primaires (primary school leaving certificate)
* free of any medical or psychiatric condition likely to interfere with cognition, other than a diagnosis of SCD / MCI
* affiliated with a social security scheme
* having received oral and written information abou the protocol and having signed a consent form to participate in this research
* patients with 'subjective cognitive decline-plus' (hereafter 'SCD', criteria of Jessen et al., 2014) or patients with mild neurocognitive impairment due to Alzheimer's disease (hereafter 'MCI', criteria of Albert et al., 2011)

Exclusion Criteria:

* contraindications to MRI : Abdominal circumference + upper limbs stuck to the body > 200 cm; Implantable pacemaker or defibrillator; Neurosurgical clips; Cochlear implants ; Neural or peripheral stimulator; Intra-orbital or encephalic metallic foreign bodies; Endoprostheses fitted less than 4 weeks ago and osteosynthesis devices fitted less than 6 weeks ago; Claustrophobia.
* sensory deficit interfering with experimental tests
* pregnant or breast-feeding women
* adults under legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty
* 7-items modified Hachinski ischemic score >2 (Hachinski et al., 2012)
* Dementia (McKhann et al., 2011)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Diffusion-MRI based parameters estimates of medial temporal lobe gray matter microstructure | 2 hours and 30 minutes
  Free-water and free-water corrected Fractional anisotropy are two parameters that can be estimated through Multi-Compartment Modelling of the diffusion MRI signal within medial temporal lobes gray matter. We will compute these parameters for the hippocampus and the surroundings rhinal cortices. These measures will be compared between patients and healthy controls.

SECONDARY OUTCOMES:
Diffusion-MRI based parameters estimates of medial temporal lobe gray matter microstructure | 2 hours and 30 minutes
  Free-water and free-water corrected Fractional anisotropy are two parameters that can be estimated through Multi-Compartment Modelling of the diffusion MRI signal within medial temporal lobes gray matter. We will compute these parameters for the hippocampus and the surroundings rhinal cortices. These measures will be compared across patients groups.
Relationships between medial temporal lobe gray matter microstructure and memory | 2 hours and 30 minutes
  Free-water and free-water corrected Fractional anisotropy are two parameters that can be estimated through Multi-Compartment Modelling of the diffusion MRI signal within medial temporal lobes gray matter. We will compute these parameters for the hippocampus and the surroundings rhinal cortices. Memory accuracy scores will be computed for the two memory tasks "The '4 mountains test' and the 'Memory entities' test" . Correlational analyses will be performed across groups between gray matter microstructure estimates and memory scores.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves JONIN, PhD, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France